CLINICAL TRIAL: NCT06363123
Title: Identification and Validation of Plasma Diagnostic Biomarkers for Multi-Cancer Based on Metabolomics: A Multi-Center Clinical Research and Validation Trial
Brief Title: Plasma Metabolic Biomarkers for Multi-Cancer Diagnosis
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Min Li, Deputy Director of Science and Technology Department, Beijing Friendship Hospital
Other Study IDs: BFHHZML20240009
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer; Breast Cancer; Colorectal Cancer; Thyroid Cancer; Gastric Cancer; Cervical Cancer; Liver Cancer; Pancreatic Cancer; Cholangiocarcinoma; Prostate Cancer; Esophageal Cancer; Ovarian Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Thyroid Neoplasms; Stomach Neoplasms; Uterine Cervical Neoplasms; Liver Neoplasms; Pancreatic Neoplasms; Cholangiocarcinoma; Prostatic Neoplasms; Esophageal Neoplasms; Ovarian Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Only metabolites will be detected and analyzed in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multi-cancer group: Patients diagnosed with cancer, including lung cancer，breast cancer，colorectal cancer，thyroid cancer，gastric cancer，cervical cancer，liver cancer，pancreatic cancer，cholangiocarcinoma，prostate cancer，esophageal cancer，ovarian cancer，renal cell carcinoma.
- control group: Healthy controls

SUMMARY:
The aim of this observational study is to comprehensively analyze the metabolites in plasma samples from multi-cancer patients using advanced mass spectrometry detection technology, in conjunction with metabolomics approaches. The goal is to construct a plasma metabolite database for multi-cancer patients. Simultaneously, we will delve into the exploration and validation of a series of metabolic biomarkers for early multi-cancer diagnosis. The objective is to establish a safer, more convenient, and more sensitive early screening method, thereby providing a reliable scientific foundation and critical evidence for improving the early diagnostic process for individuals at high risk of multi-cancer.

DETAILED DESCRIPTION:
Firstly, a wide-targeted metabolomic measurement will be conducted on all samples to identify potential metabolite candidate markers and analyze differences in the metabolic profiles of patients with different types of cancer. Additionally, a comprehensive metabolite database specific to cancer patients will be constructed.

Secondly, Samples will be randomly allocated into modeling and testing cohorts. The modeling cohort will be further divided into training and validation sets. Bioinformatics methods will be used to conduct an in-depth analysis of a wide range of metabolite information to screen out metabolic marker combinations with high diagnostic efficacy for cancer.

Ultimately, the testing cohort will be used to validate these metabolic biomarkers, aiming to ensure reliability and stability across different patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Multi-Cancer Group:

  * Patients with a confirmed diagnosis based on the clinical "gold standard".
  * Collection of plasma samples prior to treatment.
  * Availability of complete clinical data.
* Control Group:

  * Individuals with no abnormalities in routine physical examinations and relevant clinical tests.
  * Age ≥ 45 years.
  * Availability of complete clinical data.

Exclusion Criteria:

* Previous reception of anti-tumor treatments (including radiotherapy, chemotherapy, etc.) before blood collection.
* Coexistence of other systemic tumors.
* Absence of plasma sample collection before treatment.
* Pregnancy status.
* No clear evidence of histopathological diagnosis (not applicable to the control group based on this criterion).
* Patients with severe acute infections.
* Patients with severe anemia.
* Patients with severe liver or kidney dysfunction.
* Patients with autoimmune deficiency diseases.
* Patients with Hyperlipidemia.
* Patients received contrast agent injection before blood draw.
* Patients with psychiatric disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population included a range of cancer patients and healthy controls, who were admitted to the main study center and other collaborating sub-center hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Plasma metabolite content | Before receiving treatment for cancer
  The outcome will be tested by metabolomics detection technology based on mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Li Min, Ph.D., Principal Investigator — Beijing Friendship Hospital
Locations (4):
- China (4):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Hebei Tumor Hospital, Shijiazhuang, Hebei
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang